CLINICAL TRIAL: NCT03620916
Title: Comparison of the Efficacy of Postoperative Analgesia by a Single Dose of Intrathecal Morphine and Intravenous Morphine: a Randomized Trial
Brief Title: Comparison of Intrathecal and Intravenous Analgesia in Patients Undergoing Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1WB1/2018/1
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-08

CONDITIONS: Liver Diseases; Liver Cancer; Liver Metastases
Keywords: liver resection; analgesia; pain; postoperative recovery
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio into experimental and control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal morphine (Experimental): Intrathecal morphine (0,4 mg) immediately before operation
  Interventions: Procedure: Intrathecal morphine
- Intravenous morphine (Active Comparator): Intravenous morphine (0,15 mg/kg body mass) immediately after the operation
  Interventions: Procedure: Intravenous morphine

INTERVENTIONS:
Procedure: Intravenous morphine — Single dose of intravenous morphine (0,15 mg/kg body mass) immediately after the operation, patient controlled analgesia with morphine (2 mg intravenously, a least 20 min interval) over first 24 postoperative hours and subcutaneous morphine (5 mg in case of numerical rating scale>4, at least 6 hour interval) over next two days
  Arms: Intravenous morphine
Procedure: Intrathecal morphine — Single dose (0,4 mg) intrathecal morphine immediately before operation, patient-controlled analgesia with morphine (2 mg intravenously, a least 20 min interval) over first 24 postoperative hours and subcutaneous morphine (5 mg in case of numerical rating scale>4, at least 6 hour interval) over next two days in the postoperative period
  Arms: Intrathecal morphine

SUMMARY:
The aim of this prospective, interventional, randomized trial is to compare the effectiveness of postoperative analgesia using single-dose intrathecal morphine and intravenous morphine in patients undergoing liver resection. The study is to include a total 36 patients randomized in a 1:1 ratio into two groups. The study will be single-blinded with respect to outcome assessors. Patients in the experimental group (n=18) will receive a single dose (0,4 mg) intrathecal morphine immediately before operation and patient-controlled analgesia (PCA) with morphine over first 24 postoperative hours and subcutaneous morphine (5 mg in case of numerical rating scale>4) over next two days in the postoperative period. Patients in the control group (n=18) will receive a single dose of intravenous morphine (0,15 mg/kg body mass) immediately after the operation and PCA with morphine over first 24 postoperative hours and subcutaneous morphine (5 mg in case of numerical rating scale>4) over next two days. Both groups will receive antiemetic prophylaxis with dexamethasone (4 mg) and ondansetron (4 mg) and standard baseline analgesia with paracetamol (1,0 g every 6 hours) and dexketoprofen (50 mg every 8 hours). Severity of pain at rest evaluated with numerical rating scale twice daily over 3 first postoperative days will be the primary outcome measure. Secondary outcome measures will include: severity of pain at coughing evaluated with numerical rating scale twice daily over 3 first postoperative days, total dose of morphine administered with PCA, time to patient mobilization, grade of sedation, intestinal motility, solid food intake tolerance, duration of hospitalization, and postoperative complications.

DETAILED DESCRIPTION:
Effective analgesia in patients undergoing liver resection is an important measure to enhance the process of postoperative recovery. The aim of this prospective, interventional, randomized trial is to compare the effectiveness of postoperative analgesia using single-dose intrathecal morphine and intravenous morphine in patients undergoing liver resection. The study is to include a total 36 patients randomized in a 1:1 ratio into two groups. The patients scheduled for liver resection in the Department of General, Transplant and Liver Surgery (Medical University of Warsaw) will be screened for eligibility basing on inclusion and exclusion criteria. Eligible patients will be included in the study following provision of informed consent. Randomization will be performed immediately before the surgical procedure in the operating theatre. The study will be single-blinded with respect to outcome assessors. Patients in the experimental group (n=18) will receive a single dose (0,4 mg) intrathecal morphine immediately before operation and patient-controlled analgesia (PCA) with morphine over first 24 postoperative hours and subcutaneous morphine (5 mg in case of numerical rating scale>4) over next two days in the postoperative period. Patients in the control group (n=18) will receive a single dose of intravenous morphine (0,15 mg/kg body mass) immediately after the operation and PCA with morphine over first 24 postoperative hours and subcutaneous morphine (5 mg in case of numerical rating scale>4) over next two days. Both groups will receive antiemetic prophylaxis with dexamethasone (4 mg) and ondansetron (4 mg) and standard baseline analgesia with paracetamol (1,0 g every 6 hours) and dexketoprofen (50 mg every 8 hours). Severity of pain at rest evaluated with numerical rating scale twice daily over 3 first postoperative days will be the primary outcome measure. Secondary outcome measures will include: severity of pain at coughing evaluated with numerical rating scale twice daily over 3 first postoperative days, total dose of morphine administered with PCA, time to patient mobilization, grade of sedation, intestinal motility, solid food intake tolerance, duration of hospitalization, and postoperative complications. Side effects of intrathecal morphine injection and intravenous morphine administration will be monitored. The thresholds for type I and type II errors will be set at 0.05 and 0.20, respectively.

ELIGIBILITY:
Inclusion Criteria:

* liver resection
* liver malignancy

Exclusion Criteria:

* >3 points in American Society of Anesthesiology (ASA) scale
* contra-indications for intrathecal morphine administration
* chronic preoperative intake of analgetics
* a history of opioid dependency
* body mass index >45 kg/m2
* allergy to any analgetic drug administered in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Severity of pain at rest | 3 days
  Severity of pain assessed in numerical rating scale twice daily

SECONDARY OUTCOMES:
Severity of pain at coughing | 3 days
  Severity of pain assessed in numerical rating scale twice daily
Morphine usage | 3 days
  Total dose of morphine administered intravenously and subcutaneously
Time to mobilization | 90 days
  Time to self-standing after the operation
Grade of sedation | 3 days
  Richmond Agitation and Sedation Scale
Solid food tolerance | 90 days
  Time to solid food intake
Duration of hospitalization | 90 days
  Postoperative hospital stay
Postoperative complications | 90 days
  Postoperative complications according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Niewiński, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (2):
- Poland (2):
  - Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - II Department of Anaesthesiology and Intensive Care, Medical University of Warsaw, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niewinski G, Figiel W, Grat M, Dec M, Morawski M, Patkowski W, Zieniewicz K. A Comparison of Intrathecal and Intravenous Morphine for Analgesia After Hepatectomy: A Randomized Controlled Trial. World J Surg. 2020 Jul;44(7):2340-2349. doi: 10.1007/s00268-020-05437-x. PMID 32112166